CLINICAL TRIAL: NCT04543201
Title: Early Telehealth Visits for Discussion of Advanced Directives for Patients Newly Diagnosed With High Grade Glioma: Impact on Patient Care and Satisfaction
Brief Title: Telehealth Visits to Discuss Advanced Directives for Patients Newly Diagnosed With High Grade Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nimish Mohile, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UBRT21040
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early STructured Advanced care Referrals by Telehealth (Experimental): Early START visit using checklist over telephone or zoom:
  A telehealth visit conducted within 4 months of patient diagnosis, with the goal of encouraging patients to discuss and document their end-of-life wishes prior to the onset of cognitive impediments common among patients with late-stage high grade glioma.
  Interventions: Behavioral: Early START visit using checklist over telephone or zoom

INTERVENTIONS:
Behavioral: Early START visit using checklist over telephone or zoom — Prior to visit subject receives pre-visit educational guide and copy of advance directive form
  Follow up surveys:
  Immediate: provider feedback survey
  2-4 weeks after visit: subject feedback survey and caregiver/family feedback survey
  After subject death: caregiver/family survey

SUMMARY:
High grade gliomas (HGGs) are rapidly progressive brain tumors resulting in death for most patients between 6 months and 2 years after diagnosis. It is important for patients with HGG to discuss and document their wishes at the end of life. However, many of these patients experience early changes in cognition which impede their decision-making. For this reason, these patients should have early discussions with their providers. However, implementation of this remains challenging in clinical practice.

In this study, we will create an Early STructured Advanced care Referrals by Telehealth (Early START) visit for patients soon after their initial oncology visit. A checklist and pre-visit guide were developed to help guide the visit for both the provider and patient. Providers will receive special training in running these visits. Caregivers and/or family members will be encouraged to participate. Visits will be done using video or telephone and recorded. For patients who do not have access to technology for these visits, it will be provided. After the visit, patients, caregivers and/or family who participated, and providers will fill out surveys to address feasibility of having these extra visits and improve the visits for future. Patients will be followed until death. Caregivers and/or family who participated will be asked about whether end of life was in line with the patient's wishes. We will also use the patient's medical record to assess other aspects of end of life. We will compare end of life outcomes with other similar patients treated at our center.

DETAILED DESCRIPTION:
High grade gliomas (HGGs) are rapidly progressive brain tumors resulting in death for most patients between 6 months and 2 years after diagnosis. Discussion and documentation of an advance care plan are needed to achieve end of life goals that are concordant with a patient's wishes. Early cognitive dysfunction in brain tumor patients can impede patients from making decisions about their own care. Patients with HGG, therefore require discussion and documentation of end of life goals early in their disease course, but implementation of this has been elusive.

In this study, we will integrate an Early STructured Advanced care Referrals by Telehealth (Early START) visit into standard neuro-oncologic care prior to initiation of adjuvant chemotherapy in patients with HGG. Multi-disciplinary providers including physicians, advanced practice providers, and nurses will undergo an in-service by palliative care experts to perform Early START with a standardized checklist followed by periodic training sessions. Fifty patients with HGG will be enrolled over a 12-month period. They will receive a pre-visit educational guide to increase literacy regarding advance directives (AD) followed by a provider-led Early START visit that will be recorded. Post-visit assessments will address patient and caregiver perspectives on the intervention, patient and caregiver knowledge, patient satisfaction and patient-reported anxiety measures. A provider questionnaire will assess length of visit, adherence to the checklist and AD outcomes of the visit. Patients will be followed until death. End of life quality measures and concordance of death with goals of care will be assessed using a combination of caregiver surveys and the electronic medical record. These outcomes will be compared to historical controls treated at our center from 2010-2015.

Specific Aims:

Aim 1a. To determine the effectiveness of Early START as measured by AD documentation.

Aim 1b. To determine the utility of Early START as measured by timing of hospice enrollment at the end of life and place of death concordant with the patient's goals.

Hypothesis: As our primary aim, we hypothesize that Early START will increase the percentage of AD documentation by the 3rd oncology visit from 51% to 80%. As secondary outcomes, we hypothesize that it will decrease the percentage of AD that are completed by proxy from 45% to 25%, will improve end of life quality measures as compared to our published historical controls and that the majority of patients who undergo Early START will die in a setting of their choosing.

Aim 2a. To demonstrate the feasibility of Early START as measured by the percent of visits completed prior to the third oncology visit, adherence to a pre-specified checklist, and length of time to complete the visit.

Aim 2b. To optimize the Early START intervention by incorporating patient/caregiver and provider feedback.

Hypothesis: We hypothesize that 80% of visits will be completed using telehealth by the 3rd oncology visit, 80% of providers will utilize the pre-specified checklist and that average visit duration will be less than one hour.

ELIGIBILITY:
Inclusion Criteria:

* New pathologic diagnosis of WHO grade III or IV glioma within four months of consent
* English speaking

Exclusion Criteria:

* Severe cognitive dysfunction or aphasia precluding discussion of advanced care planning issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Advanced Directive Completion Rate | Time of diagnosis to 3rd oncology visit at an average of 4 months
  Percentage of patients who complete an advanced directive by the third oncology visit

SECONDARY OUTCOMES:
Early START visit completion | Time of diagnosis to 3rd oncology visit at an average of 4 months
  Percentage of Early START (Early STructured Advanced care Referrals by Telehealth) visits completed by the third oncology visit
Checklist use | Time of Early START visit [on average between 3-4 months after diagnosis]
  Percentage of providers who use the checklist
Duration of visit | Duration of visit [average 60 min]
  Duration of time in minutes
Advanced Care Directive Completion by patient vs proxy | Time of diagnosis to death up to 5 years after registration
  Percentage of completed Advanced Care Directives completed by proxy (rather than by the patient)
Chemotherapy use at end of life | Time of diagnosis to death up to 5 years after registration
  Percentage of patients that were treated with chemotherapy within 14 days of death
Hospice enrollment | Time of diagnosis to death up to 5 years after registration
  Percentage of patients who were enrolled in hospice >7 days prior to death
Palliative care and/or hospice involvement at end of life | Time of diagnosis to death up to 5 years after registration
  Percentage of patients who received a palliative care or hospice consult prior to death
Setting of end of life | Time of diagnosis to death up to 5 years after registration
  Percentage of patients for whom setting of death was consistent with their wishes

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hardy, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No